CLINICAL TRIAL: NCT05401448
Title: Study of the Non-specific Effects of Influenza and MMR Vaccine on Infectious Diseases in Goiânia, Goiás, Brazil
Brief Title: Non-specific Effects of FLU-MMR Vaccines in Adults
Acronym: FLUMMR-BRA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Faculdade da Polícia Militar, Goiânia, GO - Brazil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLUMMR-BRA
Record Dates: First submitted 2022-05-19; First posted 2022-06-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Heterologous effects of vaccines; Other viral infections
MeSH Terms: conditions — COVID-19 | interventions — Influenza Vaccines; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): sterile 0.9% NaCl
  Interventions: Other: Placebo
- Influenza (Experimental): Influenza (tetravalent vaccine)
  Interventions: Biological: Influenza
- MMR (Experimental): measles, mumps, and rubella vaccine
  Interventions: Biological: MMR vaccines

INTERVENTIONS:
Biological: Influenza — Influenza: 0.5 ml of reconstituted Influenza vaccine will be administered intramuscularly in the left upper arm as recommended by the manufacturer.
  Arms: Influenza
Biological: MMR vaccines — MMR: 0.5 ml of reconstituted MMR vaccine will be administered intramuscularly in the left upper arm as recommended by the manufacturer.
  Arms: MMR
Other: Placebo — Placebo: 0.5 ml of 0.9% NaCl will be administered intradermally in the left upper arm.
  Arms: Placebo

SUMMARY:
Various observational studies have reported an association between influenza vaccination and lower rates of infection with SARS-Cov-2 and less COVID-19 disease severity have been reported in large epidemiological studies in US, Brazil and Italy. Observational studies from the Netherlands showed also strongly reduced COVID-19 infection rates among influenza-vaccinated healthcare workers, with ORs of 0.61 and 0.49 for the first and second wave of COVID-19, respectively. In addition, in-vitro immunological analyses showed that the quadrivalent inactivated influenza vaccine can induce a trained immunity program against SARS-CoV-2 (2). In-vivo vaccination against influenza was also shown to induce improved interferon responses against SARS-CoV-2, with modulation of hyperinflammatory responses. Trained immunity could be the underlying mechanism for the potential protective effect of influenza vaccine, a mechanism that has also been proven for BCG vaccination, and epidemiological evidence suggests similar non-specific effects of MMR and OPV vaccination. Currently, various clinical trials are being conducted to study the impact of BCG, MMR and OPV vaccination on COVID-19, but prospective clinical data on influenza vaccination are lacking. Although specific COVID-19 vaccines have been developed and are proven effective, there are important reasons for assessing in a controlled randomized trial the effect of influenza and MMR vaccine on COVID19:

* Specific COVID-19 vaccines are still not yet available for all segments of the population, and especially not for the majority of the population in developing countries.
* The emergence of new SARS-CoV-2 variants, especially the P1 variant from Brazil, may very well be associated with reduced response to vaccines. An immunomodulatory protective vaccine that protects in an antigen-independent manner would be of great importance.
* It would also be conceptually important to know whether influenza and the MMR vaccine can induce heterologous protection against another viral infection, in the context of future pandemics.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, the participant must meet the following criteria:

• Be older than 18 years old. Observation: the elderly is at risk for severe forms of COVID-19, therefore, the evidence in this age group is very relevant. However, they can also be a first priority population to receive a specific vaccine, limiting the time to follow-up on the study. In addition, influenza and MMR vaccines can lead to a lower immune system in the elderly than in young people. Therefore, it is likely that a more rational choice will be to carry out the study in a young population.

Exclusion Criteria:

Participants will not be included in the study if they present (reported by the research participants):

* Known allergy to components of influenza and MMR vaccines or serious adverse events to previous administration.
* Fever (> 38 degrees Celsius) in the last 24 hours.
* Pregnancy. Note: pregnancy should be avoided for one month after vaccination.
* Symptoms of active viral or bacterial infection.
* Documented diagnosis of COVID-19.
* Vaccination in the last 4 weeks against SARS-CoV-2.
* Immunocompromised participants. This exclusion category includes: a) infection with the human immunodeficiency virus (HIV-1); b) neutropenic participant with less than 500 neutrophils/mm3; c) participant with organ transplantation; d) participants with bone marrow transplantation; e) participants in chemotherapy treatment; f) participants with primary immunodeficiency; g) participants with severe lymphopenia with less than 400 lymphocytes/mm3; h) treatment with any anti-cytokine medication; i) treatment with oral or intravenous steroids, for example, daily doses of prednisone or equivalent for more than 3 months, or probable use of oral or intravenous steroids within next four weeks.
* Some type of lymphoma or malignancy in the previous two years.
* Direct involvement in the design or execution of the study.
* Absence from work for more than 4 weeks within the next 12 weeks after study admission (vacation, maternity leave, retirement, planned surgery, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of SARS-CoV-2 infection during 1 year follow up | 3 months after inclusion
  COVID-19 will be defined as meeting the following two criteria:
  1. signs and symptoms compatible with the disease as judged by the adjudication committee based on the most recent knowledge of COVID-19
  2. microbiological or radiological confirmation: meeting any of the following: a. presence of SARS-CoV-2 virus by PCR
Cumulative incidence of SARS-CoV-2 infection | 6 months after inclusion
  COVID-19 will be defined as meeting the following two criteria:
  1. signs and symptoms compatible with the disease as judged by the adjudication committee based on the most recent knowledge of COVID-19
  2. microbiological or radiological confirmation: meeting any of the following: a. presence of SARS-CoV-2 virus by PCR
Cumulative incidence of SARS-CoV-2 infection | 12 months after inclusion
  COVID-19 will be defined as meeting the following two criteria:
  1. signs and symptoms compatible with the disease as judged by the adjudication committee based on the most recent knowledge of COVID-19
  2. microbiological or radiological confirmation: meeting any of the following: a. presence of SARS-CoV-2 virus by PCR

SECONDARY OUTCOMES:
Severity of SARS-CoV-2 and the incidence of clinically relevant RTI | 3, 6 and 12 months after inclusion
  Cumulative incidence of hospitalization for COVID-19; Cumulative incidence of ICU admission for COVID-19; Cumulative incidence of death due to COVID-19; All parameters combined, measured as number of days or number of deaths will be used to report COVID19 severity.
Severity of other respiratory tract infections (RTIs) | 3, 6 and 12 months after inclusion
  Cumulative incidence of hospitalization for other RTIs; Cumulative incidence of hospitalization for all infections; Cumulative incidence of death due to other infections;
  All parameters combined, measured as number of days or number of deaths will be used to report the severity of the infection.
  Cumulative incidence of hospitalization for all infections
Incidence and magnitude of plasma/serum antibodies (IgA, M, G) and SARS-Cov-2-specific antibodies at the end of study | 3, 6 and 12 months after inclusion
  The measurement of the antibodies titers will be used together with the self informed questionnaires in order to confirm the incidence of COVID19 and/or other RTIs.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Netea, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Faculdade da Polícia Militar, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No